CLINICAL TRIAL: NCT05848570
Title: Keeping it LITE: Exploring HIV Risk in Vulnerable Youth With Limited Interaction and Digital Health Intervention
Acronym: LITE-2
Status: Recruiting | Type: Observational
Sponsor: Hektoen Institute for Medical Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1UG3AI169631-01 (NIH)
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections; Sexual Behavior
MeSH Terms: conditions — HIV Infections; Sexual Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Keeping it LITE — observational cohort only

SUMMARY:
Despite advances in HIV diagnostics, care and prevention strategies, infection rates among adolescent and young adult sexual and gender minorities (SGM) continue to rise in the United States (US). There is an urgent need to describe the epidemiology and trajectories of HIV acquisition in this population and to offer age and culturally appropriate scalable prevention interventions to those at highest risk of infection in the US. This project will engage and retain young SGM in an innovative longitudinal cohort, enroll participants in a dynamic established digital health retention platform (HMP; HealthMPowerment), monitor HIV risk and prevention behaviors and explore the socioecological factors that influence the use of new HIV prevention technologies (UG3 phase), while also allowing targeted testing of novel digital health interventions (UH3 phase). In Aim 1, the investigators will enroll and retain a large (n=6000; 3000/year), diverse cohort of sexually active, SGM adolescents and young adults, ages 13-34, using innovative digital recruitment, engagement and retention strategies. Over the course of the study, the investigators will longitudinally characterize the sexual behavior, HIV transmission risk, and PrEP uptake trajectories of SGM youth utilizing epidemiological trajectory analyses to identify the most effective points of intervention (Aim 2). This study will capitalize upon productive existing partnerships and digital health expertise to articulate the drivers of the ongoing HIV epidemic among the most vulnerable populations in the US in order to identify the most effective, expeditious and scalable strategies to address this ongoing public health crisis.

ELIGIBILITY:
Inclusion Criteria:

* For young adults ages 18-34: self-identified SGM young adults ages 18-34 who meet at least one of the following criteria:

  * 1) condomless anal or vaginal intercourse (CAI) with a cisgender man in the last 6 months OR
  * 2) sex with cisgender men and bacterial STI in the last 6 months OR
  * 3) anal or vaginal sex with a known HIV-infected partner in the last 6 months.
* For adolescents 13-17: self-identified SGM adolescents ages 13-17 who have engaged in any sexual activity (e.g., oral, anal or vaginal sex)

Exclusion Criteria:

* under age 13
* over age 34

Ages: 13 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Self-identified sexual and gender minority adolescents and young adults ages 13-34.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Sexual Behavior Questionnaire | past 6 months
  oral, anal and vaginal sex episodes
HIV Testing Result | past 12 months
  HIV seroconversion

SECONDARY OUTCOMES:
PrEP uptake | past 6 months
  initiation of pre-exposure prophylaxis for HIV prevention

CONTACTS AND LOCATIONS:
Locations (1):
- John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided